CLINICAL TRIAL: NCT01783925
Title: Eylea Post Marketing Surveillance
Brief Title: Eylea Post Marketing Surveillance(PMS)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 16469; EY1310KR (Other: company internal)
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Patients in daily life clinical practice treatment receiving EYLEA according to indication on the label.

SUMMARY:
The objective of this PMS is to gain information about safety and efficacy in real practice as a regulatory commitment required by MFDS

ELIGIBILITY:
Inclusion Criteria:

* Patients determined to start EYLEA treatment
* Patients who agree and sign informed consent
* Patients who receive EYLEA treatment for the first time
* Patients who meet one of the following

  * Patients diagnosed by physician as having neovascular (wet) age-related macular degeneration wAMD
  * Patients diagnosed by physician as having visual impairment due to macular edema secondary to retinal vein occlusion (branch RVO or central RVO)
  * Patients diagnosed as having visual impairment due to diabetic macular edema (DME)
  * Patients diagnosed as having visual impairment due to myopic choroidal neovascularization (mCNV)

Exclusion Criteria:

* Patients who have received anti-VEGF therapy within 90 days
* Patients who are contraindicated based on the approved product label

  * Ocular or periocular infection
  * Active severe intraocular inflammation
  * Known hypersensitivity to any ingredient of this drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with wet age-related macular degeneration(wAMD), RVO, DME, and mCNV who are decided to receive EYLEA (VEGF Trap Eye) treatment
Sampling Method: Non-Probability Sample
Enrollment: 3206 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) [including serious adverse events (SAEs) and ocular AEs, especially AEs due to intravitreal injection procedure] and adverse drug reactions (ADRs) | 4 months

SECONDARY OUTCOMES:
Measurement of BCVA (prior to injection and performing other ocular assessments) by eye chart. [BCVA: Best Corrected Visual Acuity] | 4 months or 8 months
Central retinal thickness by OCT with or without.[OCT: Optical Coherence Tomography] | 4 months or 8 months
Findings of FAG and/or ICAG. [FAG: Fluorescein Angiography].ICAG: Indocyanine Green Angiography] | 4 months or 8 months
IOP(if performed, before/after injection).[IOP: Intra Ocular Pressure] | 4 months or 8 months
Measurement of fundus lesion by fundoscopy | 4 months or 8 months
Adverse events (AEs) [including serious adverse events (SAEs) and ocular AEs, especially AEs due to intravitreal injection procedure] and adverse drug reactions (ADRs) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, South Korea

REFERENCES:
- [Result] Shimura M, Fukumatsu M, Tsujimura J, Hirano K, Sunaya T; Participating Investigators. Real-World Data on Intravitreal Aflibercept for Macular Edema Secondary to Central Retinal Vein Occlusion: 24-Month Outcomes. Clin Ophthalmol. 2022 Mar 1;16:579-592. doi: 10.2147/OPTH.S344194. eCollection 2022. PMID 35256840
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/16469